CLINICAL TRIAL: NCT00000758
Title: A Phase III Randomized Trial of Topical Vaginal Fluorouracil (5-Fluorouracil, 5-FU) Maintenance Therapy Versus Observation After Standard Treatment for High-Grade Cervical Dysplasia in HIV-Infected Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Prevention
Other Study IDs: ACTG 200; 11176 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Cervix, Dysplasia
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Fluorouracil; Cervix Dysplasia; Cervix Diseases
MeSH Terms: conditions — HIV Infections; Uterine Cervical Dysplasia; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Uterine Cervical Diseases | interventions — Fluorouracil

INTERVENTIONS:
Drug: Fluorouracil

SUMMARY:
To determine the efficacy and safety of intravaginal fluorouracil administered as prophylaxis in HIV-infected women who have received standard ablative therapy (surgery) for high-grade cervical dysplasia (pre-cancer of the cervix; cervical intraepithelial neoplasia). To correlate time to recurrence of cervical dysplasia with T-cell function.

Women with HIV infection are at greater risk for cervical dysplasia. Because of the likelihood that untreated or recurrent cervical dysplasia may progress to invasive cancer, there is an urgent need to develop appropriate therapies.

DETAILED DESCRIPTION:
Women with HIV infection are at greater risk for cervical dysplasia. Because of the likelihood that untreated or recurrent cervical dysplasia may progress to invasive cancer, there is an urgent need to develop appropriate therapies.

Patients are randomized to receive either intravaginal fluorouracil or no treatment (observation only). Fluorouracil cream is self-administered via applicator at biweekly intervals for 6 months. Patients are evaluated for recurrent cervical dysplasia by cytology and colposcopy with or without biopsy.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Antiretrovirals (AZT, ddI, ddC) and immunomodulators (interferon and interleukin).
* Prophylaxis or treatment for opportunistic infections.
* Vaginal antifungal agents or other indicated vaginal medications (although not permitted on day of fluorouracil application).
* Contraceptives.
* Acyclovir (prophylaxis or treatment) in patients with a history of primary or recurrent genital herpes.

Patients must have:

* HIV infection.
* Prior cervical dysplasia (grade II or III cervical intraepithelial neoplasia) successfully treated with an ablative procedure within the past 12 weeks.
* Patients less than 18 years of age must have consent of parent or guardian.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Untreated or persistent vaginal or vulvar dysplasia.
* Colposcopy or biopsy inconclusive or positive for dysplasia.
* Active genital ulcerative disease such as syphilitic chancre or herpes ulcer.
* Adenocarcinoma in situ.

Concurrent Medication:

Excluded:

* Cytotoxic chemotherapy for malignancy.
* High-dose steroids (> 10 mg/day prednisone or its steroid equivalent).

Patients with the following prior conditions are excluded:

* Malignancy requiring cytotoxic chemotherapy within the 3 months prior to study entry.
* Prior hysterectomy.
* History of allergic reaction or severe hypersensitivity to fluorouracil.

Prior Medication:

Excluded:

* Fluorouracil (systemic or topical) within 3 months prior to study entry.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 158
Dates: Study Completion 1998-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maiman M, Study Chair; Watts DH, Study Chair
Locations (21):
- United States (19):
  - Usc La Nichd Crs, Los Angeles, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - NJ Med. School CRS, Newark, New Jersey
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (2):
  - Puerto Rico-AIDS CRS, San Juan
  - San Juan City Hosp. PR NICHD CRS, San Juan

REFERENCES:
- [Background] Robinson WR, Morris CB. Cervical neoplasia. Pathogenesis, diagnosis, and management. Hematol Oncol Clin North Am. 1996 Oct;10(5):1163-76. doi: 10.1016/s0889-8588(05)70391-9. PMID 8880203
- [Background] Maiman M, Watts DH, Andersen J. A phase three randomized trial of topical vaginal 5-fluorouracil maintenance therapy versus observation after standard treatment for high grade cervical dysplasia in HIV-infected women: ACTG 200. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:155 (abstract no 466)